CLINICAL TRIAL: NCT04505969
Title: Pilot Study to Assess Patients' and Health Workers' Needs Involved in Sickle Cell Disease Management
Brief Title: A Study Aimed to Assess the Needs of Subjects With Sickle Cell Disease and Healthcare Professionals Managing Sickle Cell Disease Patients in Selected Nigerian Centres
Status: Completed | Type: Observational
Sponsor: Fondazione per la Ricerca Farmacologica Gianni Benzi Onlus (Other)
Collaborators: Barau Dikko Teaching Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: NHREC/01/01/2007-23/03/2020
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-11

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; healthcare professionals' needs; patients'needs; questionnaires
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCD patients
  Interventions: Other: Questionnaire to assess needs
- Healthcare professionals
  Interventions: Other: Questionnaire to assess needs

INTERVENTIONS:
Other: Questionnaire to assess needs — Two questionnaires have been developed to assess the specific needs of healthcare professionals working with SCD patients and of SCD patients or parents of children with SCD

SUMMARY:
This pilot research is aimed to assess the needs of patients and health workers involved in Sickle Cell Disease (SCD) management in Nigeria. To achieve this, a questionnaire will be administered to SCD patients or parents of children affected by SCD. Another questionnaire will be administered to doctors and nurses working with SCD patients. A focus group discussion with patients/parents willing to participate will be also scheduled. Participants from the following centres will be involved: Barau Dikko Teaching Hospital Kaduna State University, Ahmadu Bello University Teaching Hospital Zaria, National Hospital Abuja, Federal Medical Centre Katsina. Data will be qualitatively and quantitatively analysed and presented as aggregated data. Consent from all the study participants will be sought. Questionnaires will be coded and no personal data will be disclosed to authorised third parties.

DETAILED DESCRIPTION:
The primary objective of this study is to understand the needs of SCD patients and health workers involved in SCD management, with particular reference to the disease management in the clinical centre. This is a descriptive, mixed method prospective questionnaire-based study.

The study is intended as a pilot experience to verify the feasibility of the action through a structured survey.

Two questionnaires have been developed: one will be administered to 30 SCD patients or parents/legally designated representatives of children affected by SCD and 30 Professionals working with SCD patients (mainly doctors and nurses) in four clinical centres in Nigeria for a total of 120 patients and 120 health workers. A focus group discussion will be run with the SCD patients/parents. Following the pilot study, a wider survey will be launched involve patients, parents and healthcare professionals in the whole country and in other centres involved in the project.

Data for this study will be collected using triangulation methods. A simple random and purposive sampling techniques will be used to select respondents for the study. The collected data for this study will be presented and analysed using SPSS and thematic analysis. The study will be conducted in four centres in Nigeria: Barau Dikko Teaching Hospital Kaduna State University (BDTH), Ahmadu Bello University Teaching Hospital Zaria (ABUTH), National Hospital Abuja (NHA), and Federal Medical Centre Katsina (FMC). The study will be performed in the framework of the "African Research and Innovative initiative for Sickle cell Education: Improving Research Capacity for Service Improvement" project (GA 824021 - ARISE - H2020-MSCA-RISE-2018).

ARISE is the EU (Horizon 2020) 4-year funded project between European, African, US and Lebanon institutions for research staff exchanges, started on 1st of January 2019. Fondazione per la Ricerca Farmacologica Gianni Benzi Onlus coordinates the ARISE project.

ELIGIBILITY:
The following inclusion criteria apply for patients/parents:

* Aged ≥ 18
* Have SCD diagnosis or having a child with a SCD diagnosis
* Attending the centre from at least 6 months
* Nigerian nationality
* Informed Consent signed

The following inclusion criteria will apply for healthcare professionals:

* Working in a SCD clinic
* At least 5 years of experience with SCD patients
* Informed Consent signed

The following exclusion criteria apply for all participants:

* Informed consent form withdrawal
* Illiterate subjects
* Any psychiatric conditions impairing the participation in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Sickle Cell Disease or parents having a child with a diagnosis of Sickle Cell Disease attending one of the clinical centres involved in the study. Healthcare professionals, e.g. doctors, nurses, working with Sickle Cell Disease patients in the clinical centres involved in the study.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Nigeria (4):
  - National Hospital Abuja, Abuja
  - Barau Dikko Teaching Hospital, Kaduna State University, Kaduna
  - Federal Medical Centre Katsina, Katsina
  - Ahmadu Bello University Teaching Hospital Zaria, Zaria

IPD SHARING:
Plan to Share IPD: Yes
The research data needed to validate the results presented in the published scientific papers will be made available for verification and re-use, unless there will arise justified reasons for keeping specific datasets confidential. This will be done in compliance with the obligation to protect results, the confidentiality obligations, the security obligations, and the obligations to protect personal data as set out in the ARISE Partnership Agreement and in the Study Protocol. All the data will be anonymised before publishing.
Time Frame: Data will be made available for verification at the time of study results publication in a peer-reviewed journal
Access Criteria: A controlled access to research data will be sought. A data access form will be made available, asking for: the purpose for data request, applicant information, brief description of the research project, description of requested data, any plan for publishing results. According to the type of data, the terms for sharing will be evaluated.

REFERENCES:
- [Background] Adewoyin AS. Management of sickle cell disease: a review for physician education in Nigeria (sub-saharan Africa). Anemia. 2015;2015:791498. doi: 10.1155/2015/791498. Epub 2015 Jan 18. PMID 25667774
- [Background] Grosse SD, Odame I, Atrash HK, Amendah DD, Piel FB, Williams TN. Sickle cell disease in Africa: a neglected cause of early childhood mortality. Am J Prev Med. 2011 Dec;41(6 Suppl 4):S398-405. doi: 10.1016/j.amepre.2011.09.013. PMID 22099364
- [Background] King L, Knight-Madden J, Reid M. Newborn screening for sickle cell disease in Jamaica: a review - past, present and future. West Indian Med J. 2014 Mar;63(2):147-50. doi: 10.7727/wimj.2013.107. Epub 2014 Apr 11. PMID 25303249
- [Background] Galadanci N, Wudil BJ, Balogun TM, Ogunrinde GO, Akinsulie A, Hasan-Hanga F, Mohammed AS, Kehinde MO, Olaniyi JA, Diaku-Akinwumi IN, Brown BJ, Adeleke S, Nnodu OE, Emodi I, Ahmed S, Osegbue AO, Akinola N, Opara HI, Adegoke SA, Aneke J, Adekile AD. Current sickle cell disease management practices in Nigeria. Int Health. 2014 Mar;6(1):23-8. doi: 10.1093/inthealth/iht022. Epub 2013 Oct 10. PMID 24114193
- [Background] Green NS, Mathur S, Kiguli S, Makani J, Fashakin V, LaRussa P, Lyimo M, Abrams EJ, Mulumba L, Mupere E. Family, Community, and Health System Considerations for Reducing the Burden of Pediatric Sickle Cell Disease in Uganda Through Newborn Screening. Glob Pediatr Health. 2016 Apr 7;3:2333794X16637767. doi: 10.1177/2333794X16637767. eCollection 2016. PMID 27336011
- [Background] Makani J, Soka D, Rwezaula S, Krag M, Mghamba J, Ramaiya K, Cox SE, Grosse SD. Health policy for sickle cell disease in Africa: experience from Tanzania on interventions to reduce under-five mortality. Trop Med Int Health. 2015 Feb;20(2):184-7. doi: 10.1111/tmi.12428. Epub 2014 Nov 17. PMID 25365928
- [Background] McGann PT, Grosse SD, Santos B, de Oliveira V, Bernardino L, Kassebaum NJ, Ware RE, Airewele GE. A Cost-Effectiveness Analysis of a Pilot Neonatal Screening Program for Sickle Cell Anemia in the Republic of Angola. J Pediatr. 2015 Dec;167(6):1314-9. doi: 10.1016/j.jpeds.2015.08.068. Epub 2015 Oct 23. PMID 26477868
- [Background] World Health Organization. Sickle-Cell Anaemia Report by the Secretariat. Fifty-Ninth World Health Assembly, c2006. Available from: http://www. apps.who.int/gb/ebwha/pdf_files/WHA59/A59_9-en.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 4 four clinical centres in Kaduna and Katsina state, Nigeria were involved in the enrollement: Barau Dikko Teaching Hospital Kaduna State University (BDTH), Ahmadu Bello University Teaching Hospital Zaria (ABUTH), National Hospital Abuja (NHA), Federal Medical Centre Katsina (FMC). Centres were selected to be easily accessible to the principal investigator and his collaborators.
  A random and purposive sampling technique was adopted. Recruitment started in August 2020 and ended in October 2020.
Groups:
- SCD Patients or Parents of Children With SCD: SCD patients or parents/legally designated representatives of children with SCD attending the selected facilities
- Healthcare Professionals Working in a SCD Clinic: Healthcare professionals working in a SCD clinic having at least 5 years of experience with SCD patients
Period: Overall Study
Arm/Group | SCD Patients or Parents of Children With SCD | Healthcare Professionals Working in a SCD Clinic
Started | 108 (After obtaining the informed consent, SCD patients, parents/legally designated representatives have been asked to complete a questionnaire. The investigator gave instructions to complete, but questionnaires were self-completed. Participants had time to complete the questionnaire in a private setting and returned completed questionnaires in a closed box, that was safeguarded by the investigators.) | 84 (After obtaining the informed consent, healthcare professionals were asked to complete a questionnaire.The investigator gave instructions, but questionnaires were self-completed. Participants had time to complete the questionnaire in a private setting and returned completed questionnaires in a closed box, that was safeguarded by the investigators. Participants received information about the time and venue for a 45-60 minutes focus group discussion, led by the study principal investigator.)
Completed | 108 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCD Patients or Parents of Children With SCD | Healthcare Professionals Working in a SCD Clinic | Total
Number analyzed (Participants) | 108 | 84 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 108 | 84 | 192
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 49 | 40 | 89
  Sex: Female | 51 | 40 | 91
  Sex: unknown | 8 | 4 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Nigeria | 108 | 84 | 192

OUTCOME MEASURES:

1. Primary Outcome: Level of Satisfaction on SCD Current Treatment and Management
Description: Likert scale from 1 (very dissatisfied) to 5 (very satisfied). This Outcome Measure was pre-specified to be measured in only SCD patients/parents.
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SCD Patients: SCD patients or parents of children with SCD
Arm/Group | SCD Patients
Number analyzed (Participants) | 106
score on a scale | 4.12 (0.76)

2. Primary Outcome: Rating of the Overall Service Quality
Description: Likert scale from 1 (very poor) to 5 (very good). This Outcome Measure was pre-specified to be measured in only SCD patients/parents.
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 103
score on a scale | 4.37 (0.62)

3. Primary Outcome: Level of Satisfaction About Nursing Care in Clinic
Description: as for outcome 1
Time Frame: Single-point, at the enrollment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 108
score on a scale | 4.22 (0.74)

4. Primary Outcome: Rating of the Facilities to Manage SCD Patients
Description: Likert scale from 1 (very poor) to 5 (very good). This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthcare Professionals: Healthcare professionals working with SCD patients
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 83
score on a scale | 4.12 (0.85)

5. Primary Outcome: Level of Satisfaction on Responsibility
Description: Healthcare professionals have been asked to indicate their satisfaction about their responsibility in the clinic, using a Likert scale from 1 (very dissatisfied) to 5 (very satisfied). This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients.
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 83
score on a scale | 4.22 (0.72)

6. Primary Outcome: Level of Global Satisfaction on the Work With SCD Patients
Description: Likert scale from 1 (very dissatisfied) to 5 (very satisfied)
Time Frame: Single-point assessment, at the enrolment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 83
score on a scale | 4.17 (0.69)

7. Secondary Outcome: Level of Appreciation of the Work
Description: Likert scale from 1 (very dissatisfied) to 5 (very satisfied). This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 84
score on a scale | 4.25 (0.73)

8. Secondary Outcome: Level of Satisfaction on Protection From Injuries and Professional Risks
Description: as for outcome 7
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 83
score on a scale | 4.00 (0.85)

9. Secondary Outcome: Level of Satisfaction on the Management of the Clinic
Description: as for outcome 7
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 83
score on a scale | 4.17 (0.69)

10. Secondary Outcome: Level of Satisfaction on the Instruction Given by Doctor About Pain Control
Description: Likert scale from 1 (very dissatisfied) to 5 (very satisfied). This Outcome Measure was pre-specified to be measured in only SCD patients or parents of children with SCD
Time Frame: Single-point assessment, at the enrollment
Population: SCD patients or parents of children with SCD
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 108
units on a scale | 4.33 (0.76)

11. Secondary Outcome: Level of Satisfaction on the Support Received at the Time of the Diagnosis
Description: as for outcome 1
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 107
units on a scale | 4.33 (0.77)

12. Secondary Outcome: Level of Satisfaction on the Involvement by Doctors in Decisions That Affect the Course of Disease
Description: as for outcome 1
Time Frame: Single-point assessment, at the enrollment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 108
units on a scale | 4.35 (0.70)

13. Secondary Outcome: Level of Satisfaction on the Services Provided in the Lab
Description: as for outcome 1
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 108
score on a scale | 4.12 (0.66)

14. Secondary Outcome: Level of Satisfaction on the Communication About Sickle Cell Disease and Its Treatment
Description: as for outcome 1
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 107
score on a scale | 4.25 (0.81)

15. Secondary Outcome: Level of Satisfaction in Communicating With Lab Technicians
Description: as for outcome 1
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 107
score on a scale | 4.07 (0.61)

16. Secondary Outcome: Level of Satisfaction in Communicating With Nurses
Description: as for outcome 1
Time Frame: Single-point assessment, at the enrollment
Population: This Outcome Measure was pre-specified to be measured in only SCD patients/parents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SCD Patients
Number analyzed (Participants) | 108
score on a scale | 4.19 (0.74)

17. Secondary Outcome: Level of Satisfaction on the Relationship You Have With the Patients
Description: as for outcome 7
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 84
units on a scale | 4.49 (0.55)

18. Secondary Outcome: Level of Satisfaction on Involvement in the Decision-making Process of Your Centre
Description: as for outcome 7
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 83
score on a scale | 4.06 (0.88)

19. Secondary Outcome: Level of Satisfaction on Professional Career Advancement
Description: as for outcome 7
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 82
score on a scale | 4.12 (0.78)

20. Secondary Outcome: Level of Satisfaction on the Decision-making Autonomy
Description: as for outcome 7
Time Frame: Single-point assessment, at the enrolment
Population: This Outcome Measure was pre-specified to be measured in only healthcare professionals working with SCD patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthcare Professionals
Number analyzed (Participants) | 82
score on a scale | 4.11 (0.94)

ADVERSE EVENTS:
Description: Information not collected, not applicable
Groups:
- Healthcare Professionals: Healthcare professionals working in a SCD clinic having at least 5 years of experience with SCD patients
Arm/Group | SCD Patients | Healthcare Professionals
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Challenges due to the COVID-19 pandemics impacted on the conduction of the study. Recruitment target was lower than expectations, timelines were extended and the protocol was amended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT04505969/Prot_000.pdf